CLINICAL TRIAL: NCT04396067
Title: Aerosol Combination Therapy of All-trans Retinoic Acid and Isotretinoin as A Novel Treatment for Inducing Neutralizing Antibodies in COVID -19 Infected Patients Better Than Vaccine : An Innovative Treatment
Acronym: Antibodies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Collaborators: New Damietta University Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Principal Investigator, New Damietta University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19
Record Dates: First submitted 2020-05-18; First posted 2020-05-20 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
Keywords: COVID 2019; Isotretinoin; Endosomal toll-like receptor 3; T Cells; IFN type1; AT1; ACE2; Alvelestat
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerosolized 13 cis retinoic acid (Active Comparator): COVID 19 infected patients will receive one dose daily of Aerosolized 13 cis retinoic acid in gradual doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  Interventions: Drug: Aerosolized 13 cis retinoic acid
- All trans retinoic acid (Active Comparator): COVID 19 infected patients will receive one dose daily of Aerosolized All trans retinoic acid in gradual doses increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled All trans retinoic acid therapy for 14 days
  Interventions: Drug: Aerosolized All trans retinoic acid
- Placebo Comparator (Placebo Comparator): 4 Placebo tablets twice daily by mouth for 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aerosolized 13 cis retinoic acid — The infected patients will receive Aerosolized 13 cis retinoic acid in gradual in one dose increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled 13 cis retinoic acid therapy for 14 days
  Arms: Aerosolized 13 cis retinoic acid
Drug: Aerosolized All trans retinoic acid — The infected patients will receive Aerosolized All trans retinoic acid in gradual one dose increases froms 0.2 mg/kg/day to 4 mg/kg/day as inhaled all trans retinoic acid therapy for 14 days
  Arms: All trans retinoic acid
Other: Placebo — Placebo is a pill or tablet that does not contain any study drug.
  Arms: Placebo Comparator

SUMMARY:
Aerosol Combination therapy of All-trans retinoic acid and Isotretinoin as A novel Treatment for Inducing Neutralizing Antibodies in COVID -19 Infected Patients better than vaccine : An innovative Treatment

Mahmoud ELkazzaz(1),Tamer Haydara(2), Mohamed Abdelaal(3), Ahmed M. Kabel(4), Abedelaziz Elsayed(5) ,Yousry Abo-amer(6) ,Hesham Attia(7)

1. Department of chemistry and biochemistry, Faculty of Science, Damietta University,Egypt.
2. Department of Internal Medicine,Faculty of Medicine, Kafrelsheikh University, Egypt
3. Department of Cardiothoracic Surgery,Faculty of Medicine, Kafrelsheikh University, Egypt
4. Department of Clinical Pharmacy, Faculty of Medicine , Tanta University,Egypt.
5. Department of Pharmaceutical Biotechnology, Faculty of Pharmacy,Tanta University,Egypt.
6. Hepatology,Gastroenterology and Infectious Diseases Department, Mahala Hepatology Teaching Hospital,Egypt
7. Department of Immunology and Parasitology, Faculty of Science, Cairo University, Egypt.

   * Study Chair ((( Dr.Tamer Hydara))), Department of Internal Medicine,Faculty of Medicine, Kafrelsheikh University, Egypt Contact: Dr.Tamer Hydara-Tel: 00201142233340 Mail: tamerhydara@yahoo.com
   * Principal Investigator ((( Mahmoud Elkazzaz))), Faculty of Science, Damietta University,GOEIC,Egypt Contact:Tel: 00201090302015 Mail: mahmoudramadan2051@yahoo.com
   * Study coordinator ((Prof/Dr Mohamed Abdelaal)), Department of Cardiothoracic Surgery,Faculty of Medicine, Kafrelsheikh University, Egypt Contact:Tel: 00201001422577 Mail: Malaal2@hotmail.com

Abstract

The pandemic of COVID-19 which is caused by severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) has infected over 20,000,000 people causing over 700,000 deaths .It has no currently approved treatments. In this clinical study we confirm that combination of isotretinoin and All trans retinoic acid can be used in the treatment of SARS-COV-2 better than vaccine according to the findings of previous studies and researches. Retenoic acid can induce neutralizing antibodies in case of corona virus (COVID-19) by restoring inhebited and exhausted T cells via inhebiting both CD13 and Angiotensin-converting enzyme-2 (ACE2). CD13 amyloid receptor which abundantly overexpressed on cell surface of lymphocyte, Dentritic cell, Macrophage, granulocytes and monocytes and is ubiquitous in respiratory tract epithelial cells, smooth muscle cells, fibroblasts, epithelial cells in the kidneys and small intestine, activated endothelial cells, and platelets In addition inhibing of Angiotensin-converting enzyme-2 (ACE2) , Angiotensin T1 protein and Angiotensin II-mediated intracellular calcium release pathway which is responsible for COVID-19 cell fusion and entry.ACE2-expressing cells are prone to SARS-CoV-2 infection as ACE2 receptor facilitates cellular viral entry and replication. A study demonestrated that patients with hypertension and diabetes mellitus may be at higher risk of SARS-CoV-2 infection, as these patients are often treated with ACE inhibitors (ACEIs) or angiotensin II type-I receptor blockers (ARBs), which have been previously suggested to increase ACE2 expression.Butisotretinoin was found to be the strongest down-regulator of ACE 2 receptors.and this will give hope for diabetic patients or patients with hypertension infected with COVID-19.Therefore we suggest that Retinoic Acid will help in inhabiting factors which may enhance antibody dependent enhancement (ADE), A phenomenon caused by covid-19 which expected to lead to failure of vaccination specially in case of corona virus (covid-19) as a hyper mutatated COVID-19 antigens can lead to (ADE) phenomenon in which IgG antibodies facilitate viral entry and fusion with infected cell through uptake of the virus-IgG complex via the Fc receptors and later viral fusion with antigen presenting cells like Dentric cells, macrophages and B cells via FcR , through the neonatal FcR instead of antibodies induced viral agglutination and this is known as antibody dependent enhancement (ADE)(2) ADE can hamper vaccine development, as a vaccine may cause the production of antibodies which, via ADE, worsen the disease the vaccine is designed to protect against. ADE in COVID-19 infection can be caused by high mutation rate of the gene that encodes spike (S) protein. In this clinical study we suggest that Hyper mutated spike protein ,lymphopenia, and impaired dentreic cells all these factors can help in and lead to delayed antibodies response and appearing after a period of covid -19 symptoms onset and this may be responsible for antibody dependent enhancement (ADE)

Keywords: COVID 2019 , Retinoic acid, Lymphopenia ,T Cells, Dentric cells , ADE, Vaccine

DETAILED DESCRIPTION:
This is a Phase 2, , randomized (1:1:1), placebo-controlled, 2-weeks, proof-of-concept study to evaluate the safety and tolerability as well as the mechanistic effect of oral administration of potent inhibitor of neutrophil elastase(Inhaled All trans retinoic acid and inhaled isotretinoin in subjects infected with COVID -19

Unfortunately, all of the vaccinated monkeys treated with the Oxford vaccine known as ChAdOx1 nCoV-19, is undergoing human trials in Britain.became infected when challenged as judged by recovery of virus genomic RNA from nasal secretions," said Dr William Haseltine, a former Harvard Medical School professor who had a pivotal role in the development of early HIV/Aids treatments. and in general future COVID-19 vaccination which depends on inactivated viral vaccine will be restricted to healthy people with strong immunity and It will not be given to patients with History of contact with a SARS-CoV-2 infection (positive in nucleic acid test). In addition to the COVID-19 viral antigens lead to stimulate antibodies formation of IgM in acute phase and IgG type in chronic phase which is facilitate viral entry and fusion with infected cell through uptake of the virus-IgG complex via the Fc family of receptors and later viral fusion with antigen presenting cells like macrophages, B cells, monocytes via FcR family, and vascular endothelium through the neonatal Fc receptor (nFcR) instead of antibodies induced viral agglutination and this is known as antibody dependent enhancement (ADE)(2).

There are various hypotheses on how ADE happens and there is a likelihood that more than one mechanism exists. In one such pathway, some cells of the immune system lack the usual receptors on their surfaces that the virus uses to gain entry, but they have Fc receptors that bind to one end of antibodies. The virus binds to the antigen-binding site at the other end, and in this way gains entry to and infects the immune cell. Dengue virus can use this mechanism to infect human macrophages, if there was a preceding infection with a different strain of the virus, causing a normally mild viral infection to become life-threatening.(3) An ongoing question in the COVID-19 pandemic is whether-and if so, to what extent-COVID-19 receives ADE from prior infection with other coronaviruses.

ADE can hamper vaccine development: ADE can hamper vaccine development, as a vaccine may cause the production of antibodies which, via ADE, worsen the disease the vaccine is designed to protect against. Vaccine candidates for Dengue virus and feline infectious peritonitis virus (a cat coronavirus) had to be stopped because they elicited ADE.(4)

ADE in coronavirus infection can be caused by high mutation rate of the gene that encodes spike (S) protein. A thorough analysis of amino acid variability in SARS-CoV-2 virus proteins, that included the S-protein, revealed that least conservative amino acids are in most exposed fragments of S-protein including receptor binding domain (RBD).(5) Delayed antibodies response and secretion after covid -19 symptoms onset is responsible for antibody dependent enhancement (ADE)

A study shows the first seroconversion day of IgA was 2 days after onset of initial symptoms, and the first seroconversion day of IgM and IgG was 5 days after onset. The positive rate of antibodies in the 183 samples was 98.9%, 93.4% and 95.1%, for IgA, IgM and IgG, respectively. The seroconversion rate for IgA, IgM or IgG was 100% 32 days after symptom onset. According to the cumulative seroconversion curve, the median conversion time for IgA, IgM and IgG was 13, 14 and 14 days, respectively. (6)

Because this immune response takes a while to show up, antibody tests will be negative for those newly infected with COVID-19, which is why they're not used for diagnosis.

"If it's the beginning of the infection, you don't pick it up, it's something that only develops later," Dr. Melanie Ott, a virologist and immunologist at the Gladstone Institutes and a professor at the University of California, San Francisco.(7)

So, the principal investigator expects that delayed antibody response and delayed immunoglobulin class switching are the main reason for antibodies infectivity and non-specificity in the highly mutated covid-19 infection

High-affinity IgG antibodies may efficiently resolve Covid -19 infection

The more than 100 COVID-19 vaccines in development mainly focus on another immune response: antibodies. These proteins are made by B cells and ideally latch onto SARS-CoV-2 and prevent it from entering cells. T cells, in contrast, thwart infections in two different ways. Helper T cells spur B cells and other immune defenders into action, whereas killer T cells target and destroy infected cells. The severity of disease can depend on the strength of these T cell responses(1).

Studies on humoral responses to infections have been mainly geared toward the production of high-affinity IgG antibodies that efficiently resolve an infection. It has been well recognised, however, that humoral immune response to infection can be a double-edged sword that either serves as a protective mechanism to resolve the infection or aggravates the tissue injury, e.g. IgG response causes fatal acute lung injury by skewing inflammation-resolving response in SARS .(8)

In the case of respiratory infection, while IgM and IgG isotypes have been the primary emphasis in characterising immunity, mucosal and systemic IgA responses that may play a critical role in the disease pathogenesis, have received much less attention.(9),(11)

High neutrophils in covid-19 infection may be the reason of delayed antibody response and severe complications

Humoral immune response, especially production of neutralizing antibody, plays a protective role by limiting infection at later phase and prevents reinfection in the future. In SARS-CoV, both T and B cell epitopes were extensively mapped for the structural proteins, S, N, M and E protein.(12) A limited serology details of SARS-CoV-2 was reported. In a preliminary study, one patient showed peak specific IgM at day 9 after disease onset and the switching to IgG by week 2.25 Interestingly, sera from 5 patients of confirmed COVID-19 show some cross-reactivity with SARS-CoV, but not other coronavirus. Furthermore, all sera from patients were able to neutralize SARS-CoV-2 in an in vitro plaque assay, suggesting a possible successful mounting of the humoral responses.(13) Whether the kinetic/titer of specific antibody correlates with disease severity remains to be investigated.(14)

In severe cases of coronavirus disease 2019 (COVID-19), viral pneumonia progresses to respiratory failure. Neutrophil extracellular traps (NETs) are extracellular webs of chromatin, microbicidal proteins, and oxidant enzymes that are released by neutrophils to contain infections. However, when not properly regulated, NETs have potential to propagate inflammation and microvascular thrombosis - including in the lungs of patients with acute respiratory distress syndrome. While elevated levels of blood neutrophils predict worse outcomes in COVID-19, the role of NETs has not been investigated. We now report that sera from patients with COVID-19 (n = 50 patients, n = 84 samples) have elevated levels of cell-free DNA, myeloperoxidase(MPO)-DNA, and citrullinated histone H3 (Cit-H3); the latter two are highly specific markers of NETs.(15)

Neutrophils Are Sophisticated Cells Able to Adapt to Changing Inflammation

Neutrophils are not simple bags of enzymes sent to kill pathogens before the adaptive immune cells move in. In fact, they are able to respond to altered inflammatory status; neutrophils can produce cytokines , alter their gene expression during inflammation and throughout "aging" and survive for significantly longer than traditionally thought, with one study placing lifespan from bone marrow at 5.4 days . As a consequence, neutrophils are able to adapt to changing conditions and direct other cells' behaviour-a task which they can perform with some sophistication.

There are a number of murine models in which the T cell responses can be exacerbated by depleting neutrophils, implying they have a regulatory role . This suppression of T cell responses by neutrophils requires close contact and development of an immunological synapse -perhaps as the mediators thought responsible, reactive oxygen species and H2O2 do not diffuse far. Uptake of apoptotic or necrotic neutrophils also inhibits DC antigen presentation and co-stimulation, resulting in reduced T cell responses-a situation which can be exploited by pathogens. For example, neutrophils capture L. major and are subsequently engulfed by DCs, suppressing antigen presentation and T cell priming

NE was also shown to inhibit maturation and function of dendritic cells, including expression of the costimulatory molecules CD40, CD80 and CD86 Inflammatory Lung Secretions Inhibit Dendritic Cell Maturation and Function via Neutrophil Elastase.(16)

Inhibitor of elastase in covid-19 infection :

1. Alvelestat was developed as treatment for lung diseases like Chronic Obstructive Pulmonary Disease. Alevelestat works by blocking certain proteins in the body that are responsible for inflammation and damage to the lungs that can lead to COPD symptoms.

   Alvelestat Inhibitor of elastase stimulate murine B lymphocyte differentiation into IgG- and IgA-producing cells via immunoglobulin class switching and inducing also known as isotype switching, isotypic commutation or class-switch recombination (CSR), is a biological mechanism that changes a B cell's production of immunoglobulin from one type to another, such as from the isotype IgM to the isotype IgG

   A study demonstrated that depletion of neutrophils improves the production of mucosal IgA and IgG after sublingual immunization with Bacillus anthracis edema toxin as adjuvant. These past studies also demonstrated that an inverse correlation exists between the number of neutrophils and production of IgA by B cells. Using specific inhibitors of elastase, we addressed whether the elastase activity of neutrophil could be the factor that interferes with production of IgA and possibly other immunoglobulin isotypes. We found that murine splenocytes and mesenteric lymph node cells cultured for 5 days in the presence of neutrophil elastase inhibitors secreted higher levels of IgG and IgA than cells cultured in the absence of inhibitors and also,This treatment however, increased the frequency of CD4+ T cells.(17) As a mucosal targeted virus, SARS-CoV-2 would be expected to generate secretory IgA (sIgA) and induce strong mucosal immunity. Indeed, the mucosal anti-viral immunity has been shown to result in part from the IgA-mediated interactions with the pathogenic microorganisms to prevent pathogens from adhering to the cell surface.(17) Upregulated IgA production may be the result of increased levels of TGF-β and IL-10 that promote antibody switching in SARS-CoV-2 infection.(17) A study reported that depletion of neutrophils before systemic injection of vaccines increased the magnitude of antigen-specific CD4+ T cell responses, and the levels of antigen-specific serum IgG responses .(18)

   Alvelestat and Sivelestat were found to stimulate AID mRNA synthesis. The NE inhibitors also induced expression of BAFF, APRIL and IL-10 mRNA in a dose-dependent manner. Neutrophil elastase and the related serine proteases cathepsin G and proteinase 3, were shown to regulate cytokine responses through activation or degradation of cytokines, cytokine receptors, or toll-like receptor .(18) This is consistent with our finding that NE inhibitors stimulate IL-10 expression, but also BAFF and APRIL in cultures of splenocytes. IL-10 was reported to regulate expression of AID for induction of Ig CSR. (19) and it is wellestablished that IL-10 facilitates Ig class switching for production of IgA (20). Thus, these data suggest that NE inhibitors stimulate antibody production through stimulation of AID and inhibition of the activation/degradation of cytokines and cytokine receptors by elastase. NE was also shown to inhibit maturation and function of dendritic cells, including expression of the costimulatory molecules CD40, CD80 and CD86 .(21). Thus, the presence of neutrophil inhibitors may have promoted the maturation of dendritic cells and their expression BAFF and APRIL and perhaps costimulatory molecules (i.e., CD40) for enhanced antibody production. Although Alvelestat and Sivelestat are specific NE inhibitors, one should consider that they might also inhibit related elastase-like enzymes. In this regard, activated human B cells were reported to express a trypsin-like serine protease on the cell surface .(22) Concluding remarks It was previously shown that neutrophil peptide defensins enhance IgG, but not IgA responses against nasally co-administered vaccine antigens .(23) Here, the study have shown that the serine protease activity of neutrophil elastase, and possibly other serine protease such as B cell elastase, also participate in the regulation of B cell biology and adaptive immunity. However, unlike neutrophil peptide defensins, NE negatively regulate differentiation of B lymphocytes into IgG and IgA secreting cells. The presence of AID generally improves antibody-based immunity.(24).

   High Neutrophils in COVID -19 infected patients are capable of causing severe damage to the lung tissue by releasing toxic proteases and reactive oxygen species if not counterbalanced by the antiproteases.
2. All-trans retinoic acid (RA) has beneficial effects when used in a variety of inflammatory skin conditions. In a study, the authors found that RA inhibited superoxide anion production and proteolytic enzyme release by human and rat neutrophils. Concomitantly, the authors found that RA-treated neutrophils were less able than untreated neutrophils to injure endothelial cells in culture even though the adhesion of the RA-treated neutrophils to endothelial cell monolayers was not diminished. Inhibition of cytotoxicity occurred over the same range of concentrations that inhibited oxygen radical formation and protease release. In additional studies, it was observed that pretreatment of endothelial cells with RA-induced resistance to subsequent injury by activated neutrophils. Finally, in vivo studies showed that pretreatment of rats for 3 days with RA (1-10 mg/day, IP) reduced the degree of injury in the lungs and skin sites after treatment with bovine serum albumin and antibodies to bovine serum albumin in the reverse-passive Arthus reaction. Thus, RA can modulate neutrophil-mediated endothelial cell injury by an effect on both the neutrophils and their target cells. Together, these effects may underlie the reduction in immune complex-mediated injury seen in experimental animals. The beneficial effects that retinoids have in a variety of inflammatory skin diseases may likewise be a reflection of their effects on the physiology of both neutrophils and endothelial cells.

Oral retinyl palmitate or retinoic acid corrects mucosal IgA responses toward an intranasal influenza virus vaccine in vitamin a deficient mice. Retinoids inhibit inflammatory TH17 T cell responses, promote regulatory T cell (Treg) responses, and regulate expression of toll-like receptors (TLRs) .(57)

So, the principal investigator expects that retinoic acid will be effective in covid -19 patients better than the other neutrophil elastase inhibitor like Alvelestat because Attia et al (2018) demonstrated that Sivelestat reduced secretion of IgM in a dose-dependent manner , IgM type of antibodies which is very important in viral neutralization and on the other hand retinoic acid stops neutrophil-mediated endothelial cell injury by an effect on both the neutrophils and their target cells.

Seconed drug is Isotretinoin(13cis RA) and ATRA may be able to inhibit COVID 2019 infection via inducing the antiviral immunity and this is discussed as follow :

A study demonstrated that 13 cis retinoic is used in treating Emphysema (emphysema is a lung condition that causes shortness of breath), Since an effective immune response against viral infections depends on the activation of cytotoxic T cells that can clear infection by killing virus-infected cells , boosting the numbers and function of T cells in COVID-19 patients is critical for successful recovery. A recent study reported that the 82.1% of COVID-19 cases displayed low circulating lymphocyte counts. A CoV infects macrophages, and then macrophages present CoV antigens to T cells. This process leads to T cell activation and differentiation, including the production of cytokines associated with the different T cell subsets (Th17), followed by a massive release of cytokines for immune response amplification. The continued production of these mediators due to viral persistence has a negative effect on NK, and CD8 T cell activation.(25)

Recent study of 522 COVID patients and 40 healthy controls from two hospitals in Wuhan, China demonstrated that T cell numbers are negatively correlated to serum IL-6, IL-10 and TNF-α concentration, with patients in decline period showing reduced IL-6, IL-10 and TNF-α concentrations and restored T cell counts. T cells from COVID-19 patients have significantly higher levels of the exhausted marker programmed cell death protein(PD-1) as compared to health controls. Moreover, increasing PD-1 and Tim-3 expression on T cells could be seen as patients progressed from prodromal to overtly symptomatic stages, further indicative of T cell exhaustion. T cell exhaustion is a progressive loss of effector function due to prolonged antigen stimulation, characteristic of chronic infections. Dendritic cell inhibition is connected to exhaustion of CD8+ T cell polyfunctionality during chronic hepatitis C virus infection. CD8 T cells produce very effective mediators to clear nCoV2019.(26)

Dendritic cells (DCs) play a key role in innate immune and adaptive immune responses. As the strongest antigen presenting cells in the organism, they effectively stimulate the activation of T lymphocytes and B lymphocytes, thus combining innate and adaptive immunity. Immature DCs have strong migration ability, and mature DCs can effectively activate T cells in the central link of startup, regulation, and maintenance of immune responses. Thus, once the maturation process of DCs is blocked, it directly affects the initiation of subsequent adaptive immune response. MERS-CoV-2 is able to affect human dendritic cells and macrophages in-vitro .Productive replication of Middle East respiratory syndrome coronavirus in monocyte-derived dendritic cells modulates innate immune response.(27)

Another study proposed that C -C chemokine receptor type 4 (CCR4) contributes to T cell lung homing imprinting. It was found that lung DCs induce the expression of CCR4 on T cells. Lung DCs-activated T cells traffic more efficiently into the lung and protect against influenza more effectively compared with T cells activated by DCs from other tissues. Lim and colleagues suggested that CXCR4 plays a role in CD8+ T cell migration to airway tissues.(28)

Dendritic cell inhibition is connected to exhaustion of CD8+ T cell polyfunctionality during chronic hepatitis C virus infection. CD8 T cells produce very effective mediators to clear nCoV2019.(29)

Presence of RA in different tissues is very imprtant for immune induction and fighting viral infection, for example, RA is present at high concentrations in the small intestine due to metabolizing dietary vitamin A by gut epithelial cells. In this local environment, RA activate and primes dendritic cells (DCs) to become CD103+ DCs that produce RA.3, 4CD103+ DCs are migratory cells that activate naive T cells in mesenteric lymph nodes to become effector T cells that contribute to both intestinal homeostasis and immunity.and also RA is an important signal that induces IgA-producing B cells. The gut homing T cells and B cells play essential roles in protecting the digestive tract from pathogens.(30) Retinoic acid (atRA) can inhibit the spontaneous apoptosis of activated human T lymphocytes in vitro. 13-cis RA activates Th2 cytokine production Enhanced circulating dendritic cell numbers.(40)

So, according to this previous studies the principal investigator suggests that T cells lymphopenia and exhaustion may be resulted by Dendritic cells (DCs) infection and inhibition by MERS-CoV-2.

Retinoic acid has profound effects on cellular proliferation and differentiation. Moreover, it has been reported that ATRA exhibits both anti-inflammatory and immunoregulatory effects. Recent studies have shown that FOXP3 expression and the immune function of Regulatory T cells (Tregs ) can be enhanced by ATRA in the immune system of both patients and mic.13Retinoic acid (RA) is produced by a number of cell types, including macrophages and dendritic cells, which express retinal dehydrogenases that convert vitamin A to its main biologically active metabolite, all-trans RA. All-trans RA binds to its nuclear retinoic acid receptors that are expressed in lymphoid cells and act as transcription factors to regulate cell homing and differentiation. RA production by CD103+ dendritic cells and alveolar macrophages functions with TGF-b to promote conversion of naive T cells into Foxp3+ regulatory T cells and, thereby, maintain mucosal tolerance.(50) So, principal investigator expects high inducing of Dendritic cells (DCs) by retinoic acid treatment which will lead to T cells activation and migration with less exhaustion phenomenon.

Researchers from Wenzhou, China looked at clinical laboratory features including lipid levels of patients with COVID 19. They found dramatic reductions in the cholesterol levels of patients infected with COVID 19, compared with healthy controls .The study provides data to suggest that cholesterol levels decline quite rapidly during the early stages of infection and increase as the patient starts to recover. Therefore, indicating that cholesterol may have an important role to play in defending the body against such infections According to our protocol depending on previous studies the principal investigator demonstrated that there is a strong relation between immune system and cholesterol levels . :-

Cellular cholesterol is a component of the plasma membrane and is also essential in cell proliferation. Regulation of intracellular cholesterol levels has been proposed as a mechanism to regulate T cell and macrophages proliferation. Intracellular cholesterol level is regulated by two competing pathways, cholesterol uptake and efflux, and ABCA1 plays a major role in the cholesterol efflux pathway. The ATRA induces ABCA1 expression and ABCA1-dependent cholesterol efflux in activated primary human CD4+ T cells implying that RA could affect T cell functions by regulating the cellular cholesterol levels.(51) ATRA upregulates ABCA1 expression only in activated CD4+ T cells, indicating that induction of ABCA1 by ATRA and 13 cis Retinoic Acid may play an important role in immune response.

Retinoic acid and liver X receptor agonist synergistically inhibit HIV infection in CD4+ T cells by up-regulating ABCA1-mediated cholesterol efflux.(52)(53)

RA also acts directly on macrophages at both mucosal sites and other immunological sites. AtRA modulates peritoneal macrophage activation by endotoxin and IFN-γ by suppressing TNF production and nitric oxide (NO) synthesis .In addition, at RA inhibits the expression of PGE2 and COX-2 and the release of TNF, which are induced by bacterial lipopolysaccharide (LPS) in murine peritoneal macrophages .(54)

A study reported recently that substance (ATRA) have preventive effects on pulmonary fibrosis by inhibiting IL-6-dependent proliferation and TGF-β1-dependent trans differentiation of lung fibroblasts. Also, another studies demonstrated that 13-cis-retinoic acid and other retinoid analogs inhibit IL-1-induced IL-6 production and that this effect is analog-specific and, at least partially, transcriptionally mediated. This effect was dose-dependent with an IC50 of 10(-7) M RA and significant inhibition being noted with doses of RA as low as 10(-8) M. IL-10 production was inhibited by ATRA administration.(55)

A study demonstrated that TLR3(-/-), TLR4(-/-), and TRAM(-/-) mice are more susceptible to SARS-CoV than wild-type mice but experience only transient weight loss with no mortality in response to infection. In contrast, mice deficient in the TLR3/TLR4 adaptor TRIF are highly susceptible to SARS-CoV infection, showing increased weight loss, mortality, reduced lung function, increased lung pathology, and higher viral titers . New studies showed that the high level of IFN-α/β produced from the TLR3-IRF3/IRF7 pathway and IFN-β is the reason for inhibiting DENV replication. 13Cis retinoic Acid induced significant upregulation of toll-like receptor 3 (TLR3) resulting in an immune response to dsRNA intermediate which can be partially generated during CoV-2 replicationTLR3 sensitized by dsRNA and cascades of signaling pathways (IRFs and NFκB activation, respectively) are activated to produce type I IFNs.(56)

.

Oral retinyl palmitate or retinoic acid corrects mucosal IgA responses toward an intranasal influenza virus vaccine in vitamin a deficient mice. Retinoids inhibit inflammatory TH17 T cell responses, promote regulatory T cell (Treg) responses, and regulate expression of toll-like receptors (TLRs) .(57) In vitro treatment of normal human monocytes with all-trans retinoic acid (ATRA) down-regulates TLR-2 expression (58), but this effect has not been examined in patients treated with systemic retinoids. Isotretinoin (13-cis retinoic acid; 13-cis RA) is the only drug capable of inducing a long-term or permanent remission of acne; however, the mechanisms leading to this durable response are unknown. Given the role of TLR-2 in initiating immune responses to P. acnes, we hypothesized that down-regulation of TLR-2 on monocytes and/or the induction of Treg responses in vivo may represent mechanisms by which isotretinoin exerts its long-term effects.

Isotretinoin(13cis RA) may be able to inhibit COVID 2019 entry via down regulation of ACE2 , AT1 protein and Ang II-mediated intracellular calcium release rather than inhibition of interleukin-6 (IL-6) and this is discussed as follow :

Many authors misunderstands the difference between ARBs, which block ATR1 receptors and the hypothesised drug that could block the COVID-19 binding site on ACE2 receptor, which is totally different from ATR1 and 2.

The COVID-19 pandemic caused by SARS-COV-2 has infected over 2,000,000 people causing over 150,000 deaths.(59) A key host cellular protein required for the virus entry is angiotensin-converting enzyme 2 (ACE2) whose expression has been demonstrated in many tissues including alveolar epithelial type II cells in lungs, oral mucosa and intestine, heart, kidney, endothelium and skin. ACE2-expressing cells can act as home cells and are prone to SARS-CoV-2 infection as ACE2 receptor facilitates cellular viral entry and replication.(60) A study demonestrated that patients with hypertension and diabetes mellitus may be at higher risk of SARS-CoV-2 infection, as these patients are often treated with ACE inhibitors (ACEIs) or angiotensin II type-I receptor blockers (ARBs), which have been previously suggested to increase ACE2 expression.(61) In another study by Sinha et al who analyzed a publicly available Connectivity Map (CMAP) dataset of pre/post transcriptomic profiles for drug treatment in cell lines for over 20,000 small molecules, isotretinoin was the strongest down-regulator of ACE 2 receptors. On the other hand, they found 6 drugs in CMAP that are currently being investigated in clinical trials for treating COVID-19 (chloroquine, thalidomide, methylprednisolone, losartan, lopinavir and ritonavir, from clinicaltrials.gov), none of which was found to significantly alter ACE2 expression (P>0.1) Moreover, another study demonstrated that isotretinoin is a Potential papain like protease (PLpro) inhibitors which is a protein encoded by SARS-CoV-2 genes and considered one of the proteins that should be targeted in COVID-19 treatment by performing target-based virtual ligand screening.As Principal Investigator discussed before that (13cRA) is the strongest down-regulator of ACE2.

The principal investigator expects that 13cRA can inhibit or dowenrgulat ACE2 by direc interaction and binding with the transmembrane ACE2, Suggesting its therapeutic potential in preventing the entry of COVID 2019 to the host cell.

Previous studies on the related severe acute respiratory syndrome coronavirus (SARS-CoV) and SARS-CoV FP FP have shown that calcium (Ca2+) plays an important role for fusogenic activity via a Ca2+ binding pocket with conserved glutamic acid (E) and aspartic acid (D) residuesdemonstrated that intracellular Ca2+ enhances MERS-CoV WT PPs infection by approximately two-fold and that E891 is a crucial residue for Ca2+interaction. Electron spin resonance revealed that this enhancement could be attributed to Ca2+ increasing MERS-CoV FP fusion-relevant membrane ordering. Intriguingly, isothermal calorimetry titration showed that MERS-CoV FP binds one Ca2+, as opposed to SARS-CoV FP which binds to two Ca2+ ion.(62)

Angiotensin II increases the intracellular calcium activity in podocytes of the intact glomerulus. The L-type Ca2+ channel blocker nicardipine did not influence the Ang II-mediated [Ca2+] increase and it has been postulated that SARS-CoV-2 binding to ACE2 may attenuate residual ACE2 activity, skewing the ACE/ACE2 balance to a state of heightened angiotensin II activity leading to pulmonary vasoconstriction and inflammatory and oxidative organ damage, which increases the risk for acute lung injury (ALI). AngII via AT1 receptors upregulates many proinflammatory genes, such as vascular cell adhesion molecule-1 (VCAM-1), intercellular adhesion molecule-1 (ICAM-1), interleukin-6 (IL-6).30 but 13cis RA specifically down-regulated the AT1 protein in a dose- and time-dependent manner. Down-regulation of the AT1 expression leads to reduced AngII-mediated intracellular calcium release Similarly with receptor down-regulation, Treatment with 13cRA resulted in a significant reduction in AT1 mRNA .(63)

Finally, the principal investigator expects that Isotretinoin will help in antibody induction against COVID-19 via inducing different types of antiviral immune factors and also, decreasing of COVID -19 hyper mutation by blocking its ACE2 receptors and preventing the virus from cell entry and replication and this will give the immune system time to recognize COVID -19.

ELIGIBILITY:
Inclusion Criteria:

Adult SARI patients with 2019-ncov infection confirmed by PCR; Absolute value of lymphocytes < 0. 6x 109/L; Severe respiratory failure within 48 hours and requires admission to ICU. (severe respiratory failure was defined as PaO2/FiO2 < 200 mmHg and was supported by positive pressure mechanical ventilation (including non-invasive and invasive mechanical ventilation, PEEP>=5cmH2O))

Exclusion Criteria:

Age < 18 Pregnant Allergic to experimental drugs and patients have the following conditions:

1. Hypercholesterolemia
2. Hypertriglyceridemia
3. Liver disease
4. Renal disease
5. Sjögren syndrome
6. Pregnancy
7. Lactation
8. Depressive disorder
9. Body mass index less than 18 points or higher than 25 points
10. Contraindications for hormonal contraception or intrauterine device.
11. Autoimmune diseases A history of organ, bone marrow or hematopoietic stem cell transplantation
12. Patients receiving anti-hcv treatment
13. Permanent blindness in one eye
14. History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery
15. The competent physician considered it inappropriate to participate in the study
16. HIV infection or other immunodeficiency or with an absolute neutrophil count ≤1.0 × 109/L
17. Abnormal liver biochemistry (alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase) >1.5 × upper limit of normal or total bilirubin > upper limit of normal (unless Gilbert's disease with normal conjugated bilirubin)
18. Any of the following laboratory abnormalities are present at baseline:

    * Platelet count <150×109/L
    * Serum albumin ≤ 3.5 g/dL
    * INR ≥1.2
    * CPK ≥ ULN.
19. Significant liver fibrosis as evidenced by Fibrosis-4 (FIB-4) score >3.25
20. History of hypersensitivity to retinoic acid or any of its excipients or the class of neutrophil elastase inhibitors Known hypersensitivity to medications used in the study procedures (e.g. midazolam, fentanyl, and lidocaine for bronchoscopy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
lung injury score | at 7 days
  Proportion of lung injury score decreased or increased after treatment

SECONDARY OUTCOMES:
Serum levels of CRP, ESR ,IL-1,IL-6,TNF and Type I interferon | at day 7 and 14 after randimization
  Serum levels of CRP, ESR ,IL-1,IL-6,TNF and Type I interferon
Serum level of COVID19 RNA | at day 7 and 14
  Serum level of COVID19 RNA
d-dimers | within 14 days
  less than 250 ng/mL, or less than 0.4 mcg/mL of blood sample
Absolute lymphocyte counts | at day 7 and 14 after randimization
  lymphocyte counts
The immune correlates of protection against future exposure to SARS-CoV-2 | within 14 days
  To determine the immune correlates of viral clearance (Antibody Titres sufficient for viral clearance and neutralizing ) against future exposure to SARS-CoV-2
Immunological profile | within 14 days
  Number of CD4 HLA-DR+ and CD38+, CD8 lymphocytes
Total duration of mechanical ventilation, ventilatory weaning and curarisation | at day 7 and 14
Occurrence of adverse event related to immunoglobulins | at day 14
  Kidney failure, hypersensitivity with cutaneous or hemodynamic manifestations, aseptic meningitis, hemolytic anemia, leuko-neutropenia, transfusion related acute lung injury (TRALI)
IgG, IgA and IgM against COVID-19 | at day 7 and 14
  serum levels of IgG and IgM against COVID-19
ACE2 expression in patients with COVID-19 infection | at day 7 and 14
  ACE2 expression in patients with COVID-19 infection
All cause mortality rate [ | at day 7 and 14
Ventilation free days | at 14 days
ICU free days | at 14 days

CONTACTS AND LOCATIONS:
Overall Officials: M.Sc. Mahmoud Elkazzaz, B.Sc of biochemistry, Principal Investigator — Damitta University; Dr.Tamer Hydara, Lecturer of Internal Medicine, Study Chair — Faculty of medicine kafr elshiekh university